CLINICAL TRIAL: NCT03246165
Title: Incidence, Predictive Factors and Complications of Delirium in Postoperative Cardiac Surgery Elderly Patients
Brief Title: Predictive Factors and Complications of Delirium
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital de Messejana (Unknown)
Responsible Party: Principal Investigator, Bruno Caramelli, Associate Professor of Cardiology, University of Sao Paulo
Other Study IDs: 825/11
Record Dates: First submitted 2017-08-07; First posted 2017-08-11 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Delirium; Surgery--Complications; Age Problem
MeSH Terms: conditions — Delirium | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cardiac surgery — Coronary bypass, heart valve replacement

SUMMARY:
The objective of this research was to determine the incidence, predisposing and triggering factors of delirium following cardiac surgery and its consequences within 30 days of surgery and during a 12-18-month follow-up in older adult patients.

DETAILED DESCRIPTION:
Delirium is a transient and fluctuating course syndrome of acute onset that is characterized by reduced level of consciousness, global cognitive dysfunction, and disorder in the sleep-wake cycle. In patients undergoing cardiac surgery, delirium is a complication that affects 2-57% of the patients, reaching as high as 73% in older subjects.

The identification of patients at high risk for delirium is important to deliver proper care and avoid the consequences of this complication. However, previous studies published on the subject have not delivered definitive results in the cardiac surgery setting. Low educational level has also been studied as a risk factor for delirium after surgery but never in a group of cardiac surgery patients that includes a significant rate of illiteracy.

The objective of this research was to determine the incidence, predisposing and triggering factors of delirium following cardiac surgery and its consequences within 30 days of surgery and during a 12-18-month follow-up in older adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiovascular surgery

Exclusion Criteria:

* Blindness,
* deafness,
* previous stroke
* dementia
* delirium at inclusion, preoperatively
* creatinine clearance < 30 ml/min
* emergency surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to perioperative evaluation for elective cardiac surgery at the hospital de Messejana in Fortaleza, Ceara.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2013-12-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Delirium | Until hospital discharge or 30 days after surgery, and for up to 18 months.
  Delirium was assessed using the Confusion Assessment Method for the Intensive Care Unit

IPD SHARING:
Plan to Share IPD: No